CLINICAL TRIAL: NCT06194968
Title: Treatment of Acute Ischemic StroKe With Intravenous UroKinase Real-world Research: a Multicenter, Prospective Study (TASK-UK)
Brief Title: Treatment of Acute Ischemic StroKe With Intravenous UroKinase Real-world Research: a Multicenter, Prospective Study
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Techpool Bio-Pharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bo Song, chief physician, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: UK-S001
Record Dates: First submitted 2023-11-10; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Urokinase-Type Plasminogen Activator; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: Urokinase
  Interventions: Drug: Urokinase
- Active Comparator: Alteplase
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Urokinase — administered intravenously
  Groups: Experimental: Urokinase
Drug: Alteplase — administered intravenously
  Groups: Active Comparator: Alteplase

SUMMARY:
The purpose of this study is to to compare the safety and effectiveness of IV urokinase with IV alteplase in the treatment of AIS in patients up to 6 hours from symptom onset.

DETAILED DESCRIPTION:
Recombinant tissue plasminogen activator (alteplase) is currently the recommended treatment of AIS in patients within 0 to 4.5 hours from symptom onset. The cost of a single treatment with this drug is around 5000 RMB (about 700 USD). In contrast, the cost of a single dose of urokinase is around 300 RMB (about 40 USD), making it much more affordable. Currently, existing evidence regarding the effectiveness and safety of urokinase is mixed. Some studies propose that urokinase thrombolysis, compared with alteplase thrombolysis, improves perfusion without increasing the incidence of adverse reactions and mortality. In some cases, using urokinase for thrombolysis even lowers the risk of systemic bleeding, comparing to alteplase. Other studies suggest that the effectiveness and safety of urokinase intreating AIS patients is infeiror comparing to alteplase . In this study, we plan to conduct a nationwide multicenter real-world study on urokinase intravenous thrombolysis with alteplase as an active control. We will observe and analyze AIS patients treated with urokinase and alteplase and compare the effectiveness, safety and economic effects. We will explore different urokinase dosage efficacy indicators and analyze relevant risk factors. This will provide data for future systematic evaluations of the clinical effects of urokinase thrombolysis which may help lower the medical costs in treating AIS while ensuring the effectiveness.

ELIGIBILITY:
Inclusion Criteria:Age: ≥18 years. Clinical diagnosis of acute ischemic stroke, defined as an event characterized by the sudden onset of an acute focal neurologic deficit, unilateral motor dysfunction or impairment of language presumed to be due to cerebral ischemia after, with imaging evidence of a causative lesion or symptoms/signs persisting for over 24 hours. CT scan should exclude hemorrhage and non-vascular etiology.

First-time occurrence or a history of stroke without significant neurological deficits (baseline mRS score ≤ 1).

Eligible for treatment with intravenous administration of urokinase or alteplase as assessed by the investigators.

Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relatives, or deferred where applicable.

-

Exclusion Criteria:Contraindications for thrombolysis (refer to the 2018 Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke, intravenous thrombolysis contraindications).

Female of childbearing potential who is known to be pregnant and/or lactating or who has a positive pregnancy test on admission.

Known history of drug (narcotics, controlled substances) abuse or addiction in the past year.

Has an expected survival of less than 90 days due to concurrent malignant tumors or severe systemic diseases Incapable to comply with the protocol due to mental illness or cognitive disorder.

Paticipants of any interventional drug or device clinical trials within 3 months prior to screening.

Unsuitable for this study in the opinion of the investigators.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke who meet all inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) 0-2 (good functional outcome) at day 90 | at day 90

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First People's Hospital of Lanzhou City, Lanzhou, Gansu
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Beiliu People's Hospital, Beiliu, Guangxi
  - Guidong People's Hospital of Guangxi zhuang Autonomous Region, Guidong, Guangxi
  - Tengxian People's Hospital, Wuzhou, Guangxi
  - Red Cross Hospital of Yulin City, Yulin, Guangxi
  - The First People's Hospital of Yulin, Yulin, Guangxi
  - Sanya People's Hospital, Sanya, Hainan
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - The People's Hospital of Anyang City, Anyang, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The Second People's Hospital of Mengjin District, Luoyang, Henan
  - Pingdingshan The Second People's Hospital, Pingdingshan, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huiji District People's Hospital, Zhengzhou, Henan
  - Affiliated Hospital of Inner Mongolia Minzu University, Tongliao, Inner Mongolia